CLINICAL TRIAL: NCT05241418
Title: Atrial Late Gadolinium Enhancement in Patients with Repaired Congenital Heart Disease
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Castellanos, Assistant Professor of Pediatrics, Boston Children's Hospital
Other Study IDs: P00040666
Record Dates: First submitted 2022-02-02; First posted 2022-02-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease; Fibrosis Myocardial; Fibrosis; Heart
Keywords: Late gadolinium enhancement; 3D late gadolinium enhancement; atrial late gadolinium enhancement; Cardiac MRI; Congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with congenital heart disease undergoing a cardiac MRI with Gadolinium: Patients with congenital heart disease who are undergoing a clinically-ordered cardiac MRI and as part of that MRI the contrast agent, Gadolinium, will be administered.
  Interventions: Diagnostic Test: Atrial 3D late gadolinium enhancement

INTERVENTIONS:
Diagnostic Test: Atrial 3D late gadolinium enhancement — We will use cardiac MRI to take a picture of the atria. This picture will be used to identify scar tissue within the atria.
  Other Names: Atrial 3D LGE

SUMMARY:
In this research study the investigators want to learn more about how well the investigators can visualize scar tissue in the heart by MRI. In patients with congenital heart disease who need a procedure in the electrophysiology laboratory, how the MRI findings match the findings in the electrophysiology laboratory is not known. This study works to answer these questions. Participants will undergo a cardiac MRI as part of the routine clinical care that was ordered by their doctors and additional imaging by cardiac MRI will be performed.

DETAILED DESCRIPTION:
Atrial arrhythmias including intra-atrial reentrant tachycardia (IART) and atrial fibrillation (AF) routinely develop after surgical repair of congenital heart disease (CHD), contributing to heart failure exacerbation, increased hospital resource use, and reduced health-related quality of life. The combination of atriotomy scars, intra-cardiac suture lines, and chronic pressure or volume overload from residual lesions creates the necessary milieu of heterogeneous atrial fibrosis capable of supporting wavefront reentry. While catheter ablation has become a primary tool in the management of IART and AF, long-term ablation outcomes have stagnated over the preceding decade despite advances in mapping and ablative technologies. Left atrial (LA) fibrosis analysis using 3-dimensional (3D) late gadolinium enhancement (LGE) cardiac magnetic resonance imaging (CMR) has shown utility in the management of adults with structurally normal hearts and atrial fibrillation (AF), having associations with endocardial bipolar voltage amplitude, likelihood of maintenance of sinus rhythm after ablation, and thromboembolic risk. Excellent reproducibility of LA fibrosis quantification has been demonstrated in adults with structurally normal hearts and AF. To date, the use of 3D LGE in CHD has been limited to the ventricles. Prior studies have described altered LA function in adolescent and young adult patients with rTOF. Additionally, right atrial (RA) functional abnormalities have also been described in patients with rTOF. No prior studies have attempted to validate this technology in the atrium of patients with congenital heart disease. Our studies aims to investigate the reproducibility of atrial fibrosis quantification by cardiac MRI and may provide insights to correlations with voltage mapping in the electrophysiology laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patients >13 years old with congenital heart disease referred for cardiac MRI and receiving gadolinium as part of routine clinical care or for pre-ablation planning will be included.

Exclusion Criteria:

* Those with self-reported anxiety or claustrophobia and/or the presence of a permanent pacemaker or implantable cardioverter defibrillator will be excluded.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The hospital at which the investigators are based is a referral center for patients with congenital heart disease. These patients sometimes require a cardiac MRI. Patients >13 years old with congenital heart disease referred for CMR and meeting eligibility criteria will be approached for this study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Total atrial fibrosis content from 3D-LGE-CMR | 1 year
  Atrial 3D-LGE-CMR images will be post-processed using the Circle ADAS 3D software module (Circle Cardiovascular Inc., Calgary, AB, Canada) and analyzed to identify fibrotic tissue. Results are portrayed as 3D-colored maps and as a calculated percentage of atrial fibrosis relative to total atrial surface area. All CMR images will be analyzed by two observers for the calculation of interrater reliability of the percent of atrial LGE. One observer will perform contours twice for the purposes of intra-observer agreement.

SECONDARY OUTCOMES:
Total atrial fibrosis content from catheter-derived endocardial bipolar voltage map. | 2 years
  In patients who have a cardiac MRI and then an electrophysiology study as part of their clinical care, the 3D-CMR image will be compared to the catheter-generated electro-anatomic voltage mapping obtained in the electrophysiology laboratory.
Sustained atrial arrhythmia, defined as IART/AF lasting >30 seconds detected on ECG, ambulatory monitor, or inpatient telemetry | 5 years
  Following 3D-LGE-CMR acquisition, CMR and clinical data will be entered into a deidentified database to be used for clinical research. After 5 years patients without a prior history of electrophysiology issues will be analyzed prospectively (over a 5 year period) for the development of a sustained atrial arrhythmia using time-to-event analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Castellanos, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouchardy J, Therrien J, Pilote L, Ionescu-Ittu R, Martucci G, Bottega N, Marelli AJ. Atrial arrhythmias in adults with congenital heart disease. Circulation. 2009 Oct 27;120(17):1679-86. doi: 10.1161/CIRCULATIONAHA.109.866319. Epub 2009 Oct 12. PMID 19822808
- [Background] Labombarda F, Hamilton R, Shohoudi A, Aboulhosn J, Broberg CS, Chaix MA, Cohen S, Cook S, Dore A, Fernandes SM, Fournier A, Kay J, Macle L, Mondesert B, Mongeon FP, Opotowsky AR, Proietti A, Rivard L, Ting J, Thibault B, Zaidi A, Khairy P; AARCC. Increasing Prevalence of Atrial Fibrillation and Permanent Atrial Arrhythmias in Congenital Heart Disease. J Am Coll Cardiol. 2017 Aug 15;70(7):857-865. doi: 10.1016/j.jacc.2017.06.034. PMID 28797355
- [Background] Akoum N, Fernandez G, Wilson B, Mcgann C, Kholmovski E, Marrouche N. Association of atrial fibrosis quantified using LGE-MRI with atrial appendage thrombus and spontaneous contrast on transesophageal echocardiography in patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2013 Oct;24(10):1104-9. doi: 10.1111/jce.12199. Epub 2013 Jul 11. PMID 23844972
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537
- [Background] Chelu MG, King JB, Kholmovski EG, Ma J, Gal P, Marashly Q, AlJuaid MA, Kaur G, Silver MA, Johnson KA, Suksaranjit P, Wilson BD, Han FT, Elvan A, Marrouche NF. Atrial Fibrosis by Late Gadolinium Enhancement Magnetic Resonance Imaging and Catheter Ablation of Atrial Fibrillation: 5-Year Follow-Up Data. J Am Heart Assoc. 2018 Dec 4;7(23):e006313. doi: 10.1161/JAHA.117.006313. PMID 30511895
- [Background] King JB, Azadani PN, Suksaranjit P, Bress AP, Witt DM, Han FT, Chelu MG, Silver MA, Biskupiak J, Wilson BD, Morris AK, Kholmovski EG, Marrouche N. Left Atrial Fibrosis and Risk of Cerebrovascular and Cardiovascular Events in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Sep 12;70(11):1311-1321. doi: 10.1016/j.jacc.2017.07.758. PMID 28882227
- [Background] Chubb H, Aziz S, Karim R, Sohns C, Razeghi O, Williams SE, Whitaker J, Harrison J, Chiribiri A, Schaeffter T, Wright M, O'Neill M, Razavi R. Optimization of late gadolinium enhancement cardiovascular magnetic resonance imaging of post-ablation atrial scar: a cross-over study. J Cardiovasc Magn Reson. 2018 May 3;20(1):30. doi: 10.1186/s12968-018-0449-8. PMID 29720202
- [Background] Rivas-Gandara N, Dos-Subira L, Francisco-Pascual J, Rodriguez-Garcia J, Pijuan-Domenech A, Benito B, Valente F, Pascual-Gonzalez G, Santos-Ortega A, Miranda B, Perez-Rodon J, Ribera-Sole A, Burcet-Rodriguez G, Roses-Noguer F, Gordon B, Rodriguez-Palomares J, Ferreira-Gonzalez I. Substrate characterization of the right ventricle in repaired tetralogy of Fallot using late enhancement cardiac magnetic resonance. Heart Rhythm. 2021 Nov;18(11):1868-1875. doi: 10.1016/j.hrthm.2021.05.032. Epub 2021 Jun 19. PMID 34098087
- [Background] Ghonim S, Ernst S, Keegan J, Giannakidis A, Spadotto V, Voges I, Smith GC, Boutsikou M, Montanaro C, Wong T, Ho SY, McCarthy KP, Shore DF, Dimopoulos K, Uebing A, Swan L, Li W, Pennell DJ, Gatzoulis MA, Babu-Narayan SV. Three-Dimensional Late Gadolinium Enhancement Cardiovascular Magnetic Resonance Predicts Inducibility of Ventricular Tachycardia in Adults With Repaired Tetralogy of Fallot. Circ Arrhythm Electrophysiol. 2020 Nov;13(11):e008321. doi: 10.1161/CIRCEP.119.008321. Epub 2020 Oct 6. PMID 33022183